CLINICAL TRIAL: NCT00065325
Title: A Randomized, Double Blind, Multicenter Study to Compare the Efficacy and Tolerability of Fulvestrant (FASLODEX™) vs. Exemestane (AROMASIN™) in Postmenopausal Women With Hormone Receptor Positive Advanced Breast Cancer With Disease Progression After Prior Non-Steroidal Aromatase Inhibitor (AI) Therapy
Brief Title: The Evaluation of the Efficacy and Tolerability of FASLODEX (Fulvestrant) and AROMASIN (Exemestane) in Hormone Receptor Positive Postmenopausal Women With Advanced Breast Cancer
Acronym: EFECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9238IL/0048; EFECT; D6997C00048
Record Dates: First submitted 2003-07-21; First posted 2003-07-23 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Locally Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: Locally advanced breast cancer; metastatic breast cancer; Breast Cancer; Cancer of Breast; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Exemestane
  Interventions: Drug: Exemestane
- 2 (Experimental): Fulvestrant
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — intramuscular injection
  Other Names: Faslodex; ZD9238
  Arms: 2
Drug: Exemestane — oral capsule
  Other Names: AROMASIN™
  Arms: 1

SUMMARY:
The purpose of this study is to compare the efficacy of Faslodex (fulvestrant) to Aromasin (exemestane) in hormone receptor positive postmenopausal women with advanced breast cancer. Patients will be treated until disease progression or until the investigator has determined that treatment is not in the best interest of the patient, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmation of Breast Cancer
* Breast Cancer has continued to grow after having received treatment with an aromatase inhibitor
* Postmenopausal women defined as a women who has stopped having menstrual periods
* Evidence of hormone sensitivity
* Written informed consent to participate in the trial

Exclusion Criteria:

* Previous treatment with Faslodex (fulvestrant) or Aromasin (exemestane)
* Any hormonal therapy used to modify the course of an additional medical condition after prior treatment with a non-steroidal aromatase inhibitor
* Treatment with an investigational or non-approved drug within one month
* An existing serious disease, illness, or condition that will prevent participation or compliance with study procedures
* A history of allergies to any active or inactive ingredients of Faslodex or Exemestane (i.e. castor oil or Mannitol)

Ages: 32 Years to 91 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2003-08; Primary Completion 2006-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Time to disease progression (TTP) | after 580 Progression events accrued

SECONDARY OUTCOMES:
Objective response rate | after 580 Progression events accrued
Overall survival | after 580 Progression events accrued
Duration of response | after 580 Progression events accrued
Clinical Benefit | after 580 Progression events accrued
Quality of Life | after 580 Progression events accrued
PK | each visit
Safety and tolerability. | after 580 Progression events accrued

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Faslodex Medical Science Director, MD, Study Director — AstraZeneca
Locations (117):
- United States (51):
  - Research Site, Birmingham, Alabama
  - Research Site, Arcadia, California
  - Research Site, Fountain Valley, California
  - Research Site, Laverne, California
  - Research Site, Long Beach, California
  - Research Site, Santa Rosa, California
  - Research Site, Torrington, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Athens, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Harvey, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Hooksett, New Hampshire
  - Research Site, Livingston, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Hershey, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Spartenburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Richmond, Virginia
- Argentina (4):
  - Research Site, Buenos Aires, Buenos Aires
  - Research Site, Ciudad de Buenos Aires, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Rosario, Santa Fe Province
- Belgium (4):
  - Research Site, Brussels, Belgium
  - Research Site, Leuven, Belgium
  - Research Site, Ottignies, Belgium
  - Research Site, Wilrijk, Belgium
- Brazil (4):
  - Research Site, Goiânia, Goiás
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
- Canada (15):
  - Research Site, Edmonton, Alberta
  - Research Site, Penticton, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, København Ø
  - Research Site, Roskilde
  - Research Site, Sønderborg
- France (4):
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Vandœuvre-lès-Nancy
- Germany (4):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Regensburg
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
- Israel (2):
  - Research Site, Haifa
  - Research Site, Tel Aviv
- Russia (3):
  - Research Site, Obninsk, Kaluga Oblast
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Africa (6):
  - Research Site, Klerksdorp, North West
  - Research Site, Bloemfontein, South Africa
  - Research Site, Cape Town, South Africa
  - Research Site, Johannesburg, South Africa
  - Research Site, Port Elizabeth, South Africa
  - Research Site, Pretoria, South Africa
- Spain (6):
  - Research Site, Seville, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, Hospitalet Dellobregat(barcelo, Catalonia
  - Research Site, Terrassa(barcelona), Catalonia
  - Research Site, Madrid, Madrid
  - Research Site, Valencia, Valencia
- Sweden (4):
  - Research Site, Halmstad
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uppsala
- Research Site, Nottingham, United Kingdom

REFERENCES:
- [Derived] Arizmendi C, Zhu Y, Khan M, Gable J, Reeve BB, King-Kallimanis B, Bell J. The FACT-GP5 as a global tolerability measure: responsiveness and robustness to missing assessments. Qual Life Res. 2024 Oct;33(10):2869-2880. doi: 10.1007/s11136-024-03740-x. Epub 2024 Jul 24. PMID 39046616
- See also: MEDLINEplus related topics: Breast Cancer — http://www.nlm.nih.gov/medlineplus/breastcancer.html
- See also: MEDLINEplus related topics: Cancer (General) — http://www.nlm.nih.gov/medlineplus/cancergeneral.html
- See also: MEDLINEplus related topics: Cancer--Living with Cancer — http://www.nlm.nih.gov/medlineplus/cancerlivingwithcancer.html
- See also: Aromasin related topics: Your Treatment with Aromasin — http://www.cancerbackup.org.uk/Treatments/Hormonaltherapies/Individualhormonaltherapies/Exemestane
- See also: CSR-9238IL-0048.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1598&filename=CSR-9238IL-0048.pdf